CLINICAL TRIAL: NCT01367106
Title: Study of the Effects in Carbohydrate Metabolism and Renal Function of "in UTERO" Exposure to Glucocorticoids in Adult Offsprings (GLUCODEX)
Brief Title: Effects of "in UTERO" Exposure to Glucocorticoids
Acronym: GLUCODEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P081209
Record Dates: First submitted 2011-05-24; First posted 2011-06-06 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: 21-hydroxylase; Defect
Keywords: offspring of 21-hydroxylase enzyme block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exposed offspring (Experimental)
  Interventions: Procedure: Euglycemic hyperinsulinemic clamp
- controls (Other)
  Interventions: Procedure: Euglycemic hyperinsulinemic clamp

INTERVENTIONS:
Procedure: Euglycemic hyperinsulinemic clamp — Euglycemic hyperinsulinemic clamp will be performed at day 2

SUMMARY:
The main objective of this study is to show that the fetal exposure to excess of glucocorticoids is associated with a deficiency of the function beta insulin in the offspring adult.

DETAILED DESCRIPTION:
The main objective of this study is to show that the fetal exposure to excess of glucocorticoids is associated with a deficiency of the function beta insulin in the offspring adult 23 subjects of exposed offspring will be compared to 23 controls

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years Aged
* Males
* Women of childbearing age with a reliable and effective contraception for over 2 months
* Taking dexamethasone between the 6th and the 24th week of gestation by the mother with bloc 21-hydroxylase or normal pregnancy for control subjects
* Normal blood pressure and heart rate measured at rest: systolic blood pressure <= 150 mmHg, diastolic blood pressure <= 90 mmHg, heart rate between 55 and 90 beats/mn.
* Normal laboratory tests or not clinically significant abnormality NFS, platelets PT, aPTT, fibrin TP, TCA, Serum electrolytes, urea, creatinine Uric acid Triglycerides, total cholesterol, HDL cholesterol
* Fating bood glucose <= 6.9 mmol/l (exclusion criteria for diabetes from the American Diabetes Association) during the OGTT.
* Negative blood HCG
* Accepting the constraints of the protocol and had signed informed and free consent.
* Affiliated to the Social Security.

Exclusion Criteria:

* Affected offspring of 21-hydroxylase enzyme block
* Taking dexamethasone until pregnancy term by the mother of the subject
* Type 2 diabetes in one of the two parents and/or 1 of the 4 grandparents
* Pregnancy, Breastfeeding
* Body Mass Index (weight/height2)> 50 kg/m2
* Poisoning smoking (>10 cigarettes per day, whatever the duration of intoxication)
* Any drug taken apart from minor analgesics (aspirin, paracetamol) for less than 8 days at the inclusion and oral contraception
* Taking recent (less than 3 months) glucocorticoids either taken orally, by inhalation or percutaneously
* Current infections or recent infections (<10 days)
* Neoplastic disorders (with the exception of carcinoma in situ of the cervix or cutaneous epithelioma), haematological, cardiovascular, psychiatric, neurological
* Having donated blood or participated in a trial within 2 months preceding their inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Glucose Tolerance | 3 days
  the tolerance will be measured by the area under the curve (AUC) of insulin secretion flow

SECONDARY OUTCOMES:
Insulin Sensitivity | 3 days
Flow measurement of insulin secretory response to intravenous glucose | 3 days
Measurement of the secretion of insulin and glucagon in response to arginine | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François GAUTIER, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Hôpital saint Louis, Paris
  - Professor GAUTIER, Paris

REFERENCES:
- [Derived] Riveline JP, Baz B, Nguewa JL, Vidal-Trecan T, Ibrahim F, Boudou P, Vicaut E, Brac de la Perriere A, Fetita S, Breant B, Blondeau B, Tardy-Guidollet V, Morel Y, Gautier JF. Exposure to Glucocorticoids in the First Part of Fetal Life is Associated with Insulin Secretory Defect in Adult Humans. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz145. doi: 10.1210/clinem/dgz145. PMID 31665349